CLINICAL TRIAL: NCT04167176
Title: Comparison of Analgesic Efficacy of Ultrasound Guided Erector Spinae Plane Block With Port Site Infiltration Following Laparoscopic Cholecystectomy
Brief Title: Comparison of Analgesic Efficacy of US Guided ESP Block With Port Site Infiltration Following Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magdy Mohammed Mahdy Sayed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABC-3-DE
Record Dates: First submitted 2019-11-06; First posted 2019-11-18 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pain
Keywords: Cholecystectomy; ESP block; Port Site Infiltration
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Active Comparator): ultrasound guided ESP Block after anaesthesia induction
  Interventions: Procedure: Erector spinae plane block; Device: Ultrasound machine (Mindray DP 9900 plus; Mindray Bio-Medical Electronics, Shenzhen, China); Drug: Bupivacaine 0.5%; Drug: Lidocaine 2%
- Port site infiltration technique (Active Comparator): After the induction of anaesthesia, pre-incisional port-site infiltration will be performed by the same surgeon every time with 20 ml of Local anesthetic (LA) mixture that will be divided equally between port sites
  Interventions: Procedure: Port site infiltration; Drug: Bupivacaine 0.5%; Drug: Lidocaine 2%

INTERVENTIONS:
Procedure: Erector spinae plane block — Patients will be placed on their right side. A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. A 21G 10-cm needle will be inserted using an in-plane approach in a cranial to caudal direction. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging. A volume of 20 mL of LA mixture (10 mL of bupivacaine 0.5%, 5 mL of lidocaine 2% and 5 mL of normal saline to make a mixture totaling 20 ml.) will be injected. The same procedure will be repeated for the opposite side.
  Other Names: ESP block
  Arms: Erector spinae plane block
Procedure: Port site infiltration — After the induction of anaesthesia, pre-incisional port-site infiltration will be performed by the same surgeon every time with 20 ml of the LA mixture. The volume will be divided equally between port sites. A total of four ports-supraumbilical, subxiphoid and two ports in the right subcostal area at mid-clavicular and anterior axillary line will be made.
  Arms: Port site infiltration technique
Device: Ultrasound machine (Mindray DP 9900 plus; Mindray Bio-Medical Electronics, Shenzhen, China) — Ultrasound will be used to identify the erector spinae muscles and to guide the LA mixture injection.
  Arms: Erector spinae plane block
Drug: Bupivacaine 0.5% — Bupivacaine 0.5% will be included in the injected LA mixture.
Drug: Lidocaine 2% — Lidocaine 2% will be included in the injected LA mixture.

SUMMARY:
To compare the efficacy of ultrasonography (USG)-guided bilateral Erector spinae plane block (ESPB) with port-site infiltration using bupivacaine for post-operative analgesia after laparoscopic cholecystectomy with a hypothesis that both Erector spinae plane block and port-site infiltration are effective in providing post-operative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* patients with the American Society of Anesthesiologists (ASA) physical status I/II,
* Age between 18 and 60 years with a body mass index (BMI) of 18-35 kg/m2,
* Patients scheduled for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Allergy to local anaesthetics,
* Infection at the site of injection,

  •, Coagulopathy,
* Chronic pain syndromes,
* Prolonged opioid medication,
* Patients who received any analgesic 24 h before surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Total postoperative opioid consumption. | 24 hours postoperatively
  Nalbuphine consumption in mg.(equivalent to morphine dose)

SECONDARY OUTCOMES:
Pain scores;Numerical Rating Scale (NRS) at rest and when coughing | at 1, 2,4 , 8, 16 and 24 hours postoperatively.
  The NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which a respondent selects a whole number (0-10 integers).
•Cumulative postoperative analgesic consumption | 24 hours postoperatively
  Analgesic drug consumption other than nalbuphine in mg.
•Heart Rate (HR) | Intraoperatively at 0, 5,10, 20, and 30 minutes. Then every 15 min thereafter till the end of surgery
  Heart Rate in beats /min
•Mean Arterial Pressure (MAP) | Intraoperatively at 0, 5,10, 20, and 30 minutes. Then every 15 min thereafter till the end of surgery
  Mean Arterial Pressure in mmHg
Incidence and severity Postoperative nausea & vomiting (PONV). | 24 hours postoperatively
  Number of patients developing PONV & PONV Score; (1) No nausea or vomiting, (2) only nausea but no vomiting, (3) single episode of vomiting or persistent nausea, and (4) two or more episodes of vomiting or severe retching.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt